CLINICAL TRIAL: NCT04359576
Title: Impact of Frozen-thawed Embryo Transfers and Hormone Substitution on Thrombotic Risk Markers
Brief Title: Frozen-thawed Embryo Transfers and Hormone Substitution on Thrombotic Risk Markers
Acronym: TromboFET
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Horsens Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Ulla Breth Knudsen, Professor, Horsens Hospital
Other Study IDs: TromboFET
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Frozen Embryo Transfer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FET: Estrogen/progesterone substituted and natural cycles
  Interventions: Diagnostic Test: Primary and secondary hemostasis

INTERVENTIONS:
Diagnostic Test: Primary and secondary hemostasis — Focus on platelet aggregation, primary and secondary hemostasis parameters

SUMMARY:
The study focus on the impact of estrogen/progesterone substitution during artificial cycle frozen embryo transfer (AC-FET) in women undertaking assisted reproductive technology treatment (ART).

DETAILED DESCRIPTION:
The aim is to investigate whether the coagulation is activated in women undergoing estrogen/progesterone substitution during artificial cycle frozen embryo transfer (AC-FET) in assisted reproductive technology treatment (ART). An activation of the coagulation might induce an increased thromboembolic risk in these women. Thus, the present study may lead to improvement of the current treatment protocol for women receiving AC-FET and ultimately prevent thromboembolic complications for woman in fertility treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women receiving FET with or without estrogen/progesterone substitution

Exclusion Criteria:

* Known bleeding disorder
* Indication for thromboprophylaxis during ART treatment
* Treatment with anti-platelet medication including non-steroid-anti-inflammatory drugs (NSAIDs) within the last week
* Donor recipients

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Healthy women receiving FET
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
coagulation | 1 year
  Primary and secondary hemostasis parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Horsens Regional Hospital, Horsens, Denmark

IPD SHARING:
Plan to Share IPD: No